CLINICAL TRIAL: NCT03397693
Title: Assessment of Endometrial Thickness & Subendometrial Perfusion by 3D Power Doppler in Women With Unexplained Infertility and PCOS.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Gadalla, Dr Moustafa Gadalla, Assistant lecturer and specialist of obstetrics and gynecology in school of medicine in Assiut University in Egypt, Assiut University
Other Study IDs: 17200152
Record Dates: First submitted 2018-01-03; First posted 2018-01-12 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Unexplained Infertility; PCOS; Endometrial Thickness
Keywords: PCOS; Unexplained infertiltiy; 3D Power Doppler; Endometrial thickness; Subendometrial blood perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Women with unexplained infertiltiy with no treatment given
- 2: Women with Poly Cystic Ovary Syndrome (PCOS) who are not being treated with drugs of ovulation induction.
- 3: Control fertile women with no treatment given.

SUMMARY:
Evaluation of the endometrial thickness and subendometrial blood perfusion in women with unexplained infertility and PCOS using 3D Power Doppler and uterine artery Doppler in comparison to a control group.

DETAILED DESCRIPTION:
• Background Infertility is a frustrating disease that affects many couples around the world. Although there are many etiologies responsible for infertility , there are about 15-30 % of couples who suffer from what is called "Unexplained Infertility". About 25% of infertility is caused by ovulatory disorders. The World Health Organization (WHO) classifies these ovulatory disorders into 3 groups. Group II includes women with hypothalamic-pituitary-ovarian dysfunction (predominately polycystic ovary syndrome (PCOS)) In unexplained infertility, basic investigations that are done first to reveal the cause of infertility reveal normal findings. These basic investigations should provide evidence of ovulation, adequate sperm production and patency of the fallopian tubes.

However, with these routine investigations and even with other more sophisticated investigations it is hard to reveal all possible abnormalities. Therefore, unexplained infertility appears to represent either the lower extreme of the normal distribution of fertility, or it arises from a defect in fecundity that cannot be detected by the routine infertility evaluation. Couples with unexplained infertility suffer from both diminished and delayed fecundity.

Due to absence of specific abnormality in cases with unexplained infertility, the management is usually empiric. Suggested treatment regimens include intrauterine insemination (IUI), ovulation induction with oral or injectable medications, combination of IUI with ovulation induction, and assisted reproductive technologies (ART).

Polycystic ovary syndrome (PCOS) is the most common endocrine disorder affecting young women of reproductive age with the prevalence ranging between 2% to 18% according to different population and diagnostic criteria. It has been suggested that uterine blood flow is impaired in women with PCOS.

Ovulation induction (OI) is by far the most commonly used treatment for women with WHO group II anovulation and clomiphene citrate (CC) has historically been the most used drug In many fertility guidelines, CC is recommended as the first-line treatment for women with group II anovulation or PCOS who wish to conceive. However, other guidelines recommend both CC and letrozole as first-line treatments. It is hypothesized that CC resistance and failure are related to anti-estrogenic effects of CC on the endometrium, cervical mucus, and uterine blood flow.

Each month, the human endometrium undergoes a series of distinct cyclical changes in preparation to receive the developing blastocyst. Such changes necessitate well-controlled dynamic remodeling of the endometrial microvasculature through the processes of angiogenesis and arteriogenesis. Abnormalities of endometrial blood perfusion have been associated with several menstrual disorders including: dysmenorrhea, menorrhagia, intermenstrual bleeding and endometriosis. So, adequate blood perfusion of the endometrium is considered an important factor for what is called "endometrial receptivity". So it is possible that women with unexplained infertility have decreased uterine and endometrial blood perfusion.

Following implantation, there are certain changes that occur in the endometrium and its vasculature. These changes occur simultaneously with the trophoblastic invasion of the spiral arteries, and any kind of abnormalities in these changes has been associated with complications during pregnancy like: recurrent miscarriage, preterm delivery, intrauterine growth restriction and pre-eclampsia. So, the condition of the endometrium is very essential for successful implantation of the gestational sac and one of the most important factors affecting the endometrium is its blood perfusion.

The usual methods of assessment of endometrium like measurement of its thickness and description of its appearance are considered poor indicators of successful implantation and pregnancy.Other tools of investigations include: uterine artery Doppler and pulsed wave Doppler. It was found that information revealed from uterine artery Doppler alone may not represent the perfusion of the endometrium. Also, pulsed wave Doppler is used to examine the smaller downstream radial and spiral arteries and this reveals information from single vessels rather than from the endometrium as a whole. On the other hand, 3D Power Doppler is claimed to be the best investigatory tool for the study of endometrial blood perfusion as it is more sensitive to low flow and thus overcomes the problems of angle dependence and background noise associated with both color and pulsed wave Doppler. In addition, whereas color Doppler provides qualitative information, the 3D Power Doppler signal can be subsequently analyzed to produce quantitative information through one of several computer software packages.

• Hypothesis: Null hypothesis: There is no difference in endometrial thickness, 2D and 3D Power Doppler indices between normal fertile women, women with unexplained infertility and women with PCOS.

Alternative hypothesis: There is a difference in endometrial thickness, 2D and 3D Power Doppler indices between above-mentioned groups.

ELIGIBILITY:
Inclusion Criteria:

* • Inclusion criteria of study group (1&2):

  1. Women with primary or secondary infertility for more than 1 year due to unexplained infertility (normal regular menstrual cycles and normal pelvic examination, evidence of ovulation by TV/US and/or normal mid-luteal serum progesterone, normal semen analysis of the husband according to WHO guidlines2010 (25), and evidence of tubal patency and normal uterine cavity by HSG and/or laparoscopy).
  2. Women with PCOS according to Rotterdam ASRM/ESHRE criteria(26) • Inclusion criteria for control group (2):

  <!-- -->

  1. Women with no history of menstrual dysfunction or subfertility.
  2. Normal regular cycles and normal pelvic examination.
  3. Multipara with last delivery since ≥ 2 years with no history of abortions and not on contraception (hormonal or IUD).

Exclusion Criteria:

* • Exclusion criteria of both groups:

  1. History of pelvic surgery or pelvic inflammatory disease.
  2. Current hormonal contraception.
  3. On IUD.
  4. History of or clinical features suggesting endometriosis or pelvic pathology like uterine fibroid and ovarian cyst.
  5. General medical disorders (e.g. D.M), smoking and lactation.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: 1. unexplained infertility (normal regular menstrual cycles and normal pelvic examination, evidence of ovulation by TV/US and normal mid-luteal serum progesterone, normal semen analysis of the husband according to WHO guidlines2010 (25), and evidence of tubal patency and normal uterine cavity by HSG and/or laparoscopy).
  2. Women with PCOS according to Rotterdam ASRM/ESHRE criteria(26)
  3. Healthy fertile women (Multipara with last delivery since ≥ 2 years with no history of abortions and not on contraception (hormonal or IUD)).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  Thickest part of the endometrium in sagittal plane by transvaginal ultrasound
Endometrial and sub-endometrial blood perfusion expressed as VI, FI VFI. | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  Endometrial and sub-endometrial blood perfusion by 3D Power Doppler
2D Doppler indices of both uterine arteries | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  RI, PI of uterine arteries.

SECONDARY OUTCOMES:
Demographic characteristics of included women. | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  Demographic characteristics of included women.
Endometrial volume | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  Using VOCAL software during transvaginal ultrasound examination
Uterine volume | Mid luteal phase defined as (Day 20-24) of the menstrual cycle for each patient
  Using VOCAL software during transvaginal ultrasound examination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, School of Medicine, Assiut University, Asyut, Egypt